CLINICAL TRIAL: NCT00490282
Title: A Pilot Trial of Image-Guided Adaptive Radiotherapy for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-0947; NCI-2012-02092 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Head and Neck Cancer; Oropharyngeal Cancer
Keywords: Head and Neck Cancer; Oropharyngeal Cancer; Adaptive Radiotherapy; Intensity Modulated Radiation Therapy; IMRT; ART
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Image-Guided Adaptive Radiotherapy (Experimental): Intensity Modulated Radiotherapy (IMRT) + Adaptive Radiotherapy (ART)
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Radiation: Adaptive Radiotherapy

INTERVENTIONS:
Radiation: Intensity Modulated Radiation Therapy — IMRT Treatment Over 6-7 Weeks
  Other Names: IMRT
Radiation: Adaptive Radiotherapy — ART Treatment Over 6-7 Weeks
  Other Names: ART

SUMMARY:
The goal of this clinical research study is to use computed tomography (CT) scans to measure and guide your radiation therapy. Researchers want to learn if the CT scans can be used to adapt radiation therapy to the changes in normal tissue and to the shrinking of the tumor that may occur as a reaction to radiation therapy. Researchers also want to see if magnetic resonance imaging (MRI) scanning can detect certain changes in the tumor any earlier than with standard tests.

DETAILED DESCRIPTION:
The Study Scans and Tests:

IMRT is a type of 3-dimensional (3-D) radiation therapy that can focus radiation beams directly on the tumor itself. In this study, the IMRT is given using a standard radiation machine (ExaCT™ machine) that has a CT scanner attached to it. This machine is commonly used in patients with head and neck cancer. It gives the same radiation treatment as most of the other machines at M. D. Anderson. However, in addition to giving radiation treatments, it can also perform CT scans while the patient is in the same position on the treatment table, before the radiation therapy is given.

For this study, your standard of care daily CT scans will be used to help researchers adjust participants' radiation therapy, if necessary, on a weekly basis. In particular, the changes in normal tissue that are being studied are any changes in the salivary glands. An additional research related MRI scan will also be performed in this study, but the MRI scan will not be used to adjust participants' therapy. Researchers want to learn if MRI scanning may be able to help doctors in the future to adjust someone's treatment based on changes in a tumor (its features and size) in response to radiation.

Enrollment in the Study:

If you agree to take part in this study, you will receive IMRT according to the standard schedule (over 6 - 7 weeks). You will sign a separate consent form for the IMRT, and the procedure and its risks will be explained to you at that time.

CT Scans:

During this study, you will have a standard of care CT scan right before each IMRT treatment (over a 6-7 week period of time, depending on the exact schedule your doctor decides would be best for your treatment). These CT scans are standard of care, are used to make sure your treatment is being aimed properly, and would be performed whether you are participating on this trial or not. Once you are set up on the treatment table and are ready for radiation therapy, the table will be turned around and the CT scan will be performed. After the CT scan, which should take about 5-8 minutes, the table will be turned back around to the original position and the radiation treatment will be given to you. In total, about 30-33 CT scans will be performed for this study, depending on the exact number of treatments the doctor decides would be best for your therapy.

Routine MRI Scans:

Routine MRI scans of your head and neck will be performed before treatment (at Week 1) and after treatment (sometime during Weeks 12-14). These scans may be used for routine treatment planning and checking the status of the disease.

Study-Related MRI Scan:

An additional MRI scan will be done halfway through treatment (during Week 3). This MRI scan will be used to help researchers see if MRI scanning may be able to help doctors in the future to adjust someone's treatment based on changes in a tumor (its features and size) in response to radiation. In 15 participants, a repeat baseline study-related MRI scan will be done 48 hours to 1 week following the first routine MRI scan.

Modified Barium Swallow:

Your swallowing function will be tested with a special type of x-ray called a modified barium swallow (MBS). During the test, you will eat and drink foods and liquids mixed with a "contrast" chemical called barium that will make your throat more visible in the x-rays. A special x-ray tube will be connected to a television screen to allow the doctor to watch the foods and liquids pass from your mouth and down your throat.

MBS will be performed before you start radiation therapy, 4-6 months after the end of radiation therapy, and during your routine follow-up visits, 12 months (plus or minus 2 months), and 24 months (plus or minus 3 months).

Saliva Testing:

One reason IMRT is being used is to try to protect your parotid glands (the largest of the salivary glands) from receiving too much radiation. To check this, a study-related saliva test will be done. For this test, the amount of saliva your parotid glands create will be measured before treatment (within 7 days before Week 1) and at the last week of treatment (during Week 6 or 7). Do not eat or drink anything, or put anything in your mouth, for 1 hour before the saliva collections. You will be asked to let your saliva collect in your mouth for 5 minutes and then spit into a cup. After that, you will be given a mild citric acid solution (like lemon juice) to put in your mouth. You will let the saliva collect in your mouth for 5 minutes and then spit in a cup. Saliva testing will be performed under a separate protocol (LAB07-0050).

Length of Study:

If the disease gets worse or intolerable side effects occur, you will be taken off this study.

Follow-Up Visits:

At some time between Weeks 22 and 24, then every 3-4 months for up to 2 years after the last IMRT, you will return for follow-up visits. The amount of saliva your parotid glands create will be measured 6 weeks after radiation therapy, 4-6 months after radiation therapy, 1 year (plus or minus 2 months) after radiation therapy, and 2 years (plus or minus 3 months) after radiation therapy.

This is an investigational study. The ExaCT™ machine is FDA approved for use in IMRT in patients with head and neck cancer. Researchers are using this standard of care CT Scan for routine quality assurance to make sure your treatment is given correctly. Up to 45 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years of age with histologically proven squamous cell carcinoma of the oropharynx, dispositioned to receive definitive radiotherapy for intact primary tumor.
2. Stage III, IVa, or IVb disease as defined by American Joint Committee on Cancer (AJCC) cancer staging criteria.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Exclusion Criteria:

1. Patients who have undergone definitive resection of the primary tumor.
2. Prior cancer diagnosis, except appropriately treated localized epithelial skin cancer or cervical cancer.
3. Prior radiation therapy to the head and neck region.
4. Patients unable or unwilling to give written, informed consent or to undergo MRI imaging.
5. Women of childbearing potential (A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 consecutive months]) and male participants must practice effective contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study
6. Patients unable to tolerate DW-MRI or DCE-MRI or having an estimated glomerular filtration rate (GFR) < 60 ml/min/1.73m2.
7. Patients who have had prior chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Garden, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 20, 2007 to November 09, 2010. All recruitment was done at The University of Texas (UT) MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Image-Guided Adaptive Radiotherapy
Started | 25
Completed | 22
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Image-Guided Adaptive Radiotherapy
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 54 [38 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Dosimetric Comparisons With Adaptive Radiotherapy (ART) Planning to Intensity-modulated Radiation Therapy (IMRT) Planning
Description: Comparison of mean dose in the Contralateral Parotid Gland and Ipsilateral Parotid Gland change between one adaptive replan (ART1) and two adaptive replans (ART2) planning relative to standard intensity-modulated radiation therapy (IMRT) planning. Dosimetric comparisons was performed using paired t-testing between plans, with patients serving as their own controls. The median trigger point for ART1 was the 16th treatment fraction. For ART2 patients, the median trigger points for the first and second replanning were the 11th and the 22nd fractions, respectively. Percent change in mean dose calculated for each group as 100% (mean post baseline (ART1 or ART2) dosage minus mean baseline IMRT dose for each parotid gland
Time Frame: Baseline by IMRT plan and adaptive dosing by ART plan evaluated during a 6-7 week course of treatment
Population: All patients had an original IMRT plan (22) and then either ART 1 (14) or ART2(8) ; Art1 and ART2 were then comparisons of the each ART with the original IMRT. The Measure type Number represents the actual percentage mean dose reduction from the comparison of mean dose in the Contralateral Parotid Gland and Ipsilateral Parotid Gland change between one adaptive replan (ART1) and two adaptive replans (ART2) planning relative to standard intensity-modulated radiation therapy (IMRT) planning.
Measure: Number; unit: percentage in mean dose reduction
Groups:
- ART1: Intensity Modulated Radiotherapy (IMRT) + IGRT with one adaptive replan (ART1)
  Intensity Modulated Radiation Therapy: IMRT Treatment Over 6-7 Weeks
  Adaptive Radiotherapy: ART Treatment Over 6-7 Weeks
- ART2: Intensity Modulated Radiotherapy (IMRT) + IGRT with two adaptive replans (ART2)
  Intensity Modulated Radiation Therapy: IMRT Treatment Over 6-7 Weeks
  Adaptive Radiotherapy: ART Treatment Over 6-7 Weeks
Arm/Group | ART1 | ART2
Number analyzed (Participants) | 14 | 8
percentage in mean dose reduction
  Contralateral Parotid Gland | -2.8 | -3.8
  Ipsilateral Parotid Gland | -3.9 | -9

2. Secondary Outcome: Number of Participants With Overall Shrinkage of Tumor With Adaptive Radiotherapy (ART)
Description: Measure parotid volumes shrinkage for the first adaptive radiotherapy (ART1) replanning for the number of participants at the median trigger point of 16th treatment fraction.
Time Frame: Baseline by IMRT plan and adaptive dosing by ART plan evaluated at the end of the 6-7 week course of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | ART1
Number analyzed (Participants) | 22
Participants | 15

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during weekly visit from baseline to ART, up to 7 weeks.
Arm/Group | Image-Guided Adaptive Radiotherapy
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes